CLINICAL TRIAL: NCT04948372
Title: Effects of Terlipressin Added to Usual Care vs. Usual Care Alone on Renal Perfusion in Patients With Septic Shock
Brief Title: Effects of Terlipressin on Renal Perfusion in Patients With Septic Shock
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, Clinical Professor, Southeast University, China
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019ZDSYLL196-P01
Record Dates: First submitted 2021-05-26; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Septic Shock
Keywords: septic shock; terlipressin; renal perfusion; acute kidney injury
MeSH Terms: conditions — Shock, Septic; Acute Kidney Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The terlipressin group (Experimental): Patients in the terlipressin group received a fixed dose of terlipressin added to usual care. Terlipressin was intravenously pumped at a fixed dose of 1.3μg/kg/hour for 24 hours.
  Interventions: Drug: Terlipressin treatment
- The usual care group (Placebo Comparator): Patients in the usual care group were treated with standard care.
  Interventions: Drug: Usual care

INTERVENTIONS:
Drug: Terlipressin treatment — Patients in the terlipressin group received a fixed dose of terlipressin added to usual care. Terlipressin was intravenously pumped at a fixed dose of 1.3μg/kg/hour for 24 hours.
  Arms: The terlipressin group
Drug: Usual care — Patients in the usual care group were treated with standard care, according to the international guidelines for the management of sepsis and septic shock.
  Arms: The usual care group

SUMMARY:
This open-label, randomized controlled trial aimed to investigate the effect of a fixed dose of terlipressin added to usual care vs. usual care alone on renal perfusion in patients with septic shock.

DETAILED DESCRIPTION:
Terlipressin is a synthetic vasopressin analog with great affinity to the V1 receptor (vasoconstrictive effect), and could selectively contract efferent arterioles, increase glomerular filtration pressure and renal perfusion. The investigators conducted this open-label, randomized controlled trial to observe the effects of a fixed dose of terlipressin added to usual care vs. usual care alone on renal perfusion in patients with septic shock. Renal perfusion was monitored by renal contrast-enhanced ultrasound. The primary outcome was peak intensity (renal perfusion parameter) at 24 hours after enrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult septic shock patients (age≥18 years old)
2. Norepinephrine dose was more than or equal to 15μg/min

Exclusion Criteria:

1. Age older than 85 years
2. Serum creatinine more than 177 μmol/L
3. Acute myocardial ischemia
4. Acute mesenteric artery ischemia
5. Pregnancy
6. Expected death within 24 hours.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2020-05-31 (Actual); Study Completion 2020-06-28 (Actual)

PRIMARY OUTCOMES:
Peak intensity | 24 hours after enrollment
  Peak intensity is the peak concentration of contrast agent, a kind of renal perfusion parameter monitored by renal contrast-enhanced ultrasound.

SECONDARY OUTCOMES:
urine output, mL | 24 hours after enrollment
  urine output with 24 hours
The incidence of acute kidney injury | Within 28 days
  Defined as serum creatinine increase≥50% within seven days or increase≥26.5 μmol/L within 48 hours

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No